CLINICAL TRIAL: NCT05694728
Title: A Phase II Trial in Healthy Chinese Women Ages 20-45 to Evaluate the Immunogenicity and Safety Profile of Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli)
Brief Title: A Phase II Trial Evaluate the Immunogenicity and Safety Profile of HPV Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Health Guard Biotechnology, Inc (Industry)
Collaborators: Jiangsu Province Centers for Disease Control and Prevention (Network); National Institutes for Food and Drug Control, China (Other); Nanjing Sangruisi pharmtech Ltd. (Unknown); Shanghai Canming pharmtech Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLWS-V502-02
Record Dates: First submitted 2022-12-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-12

CONDITIONS: Human Papilloma Virus Infection
Keywords: CIN; VIN; VaIN; AIN; Cervical cancer; Vulvar cancer; Anal cancer; Genital warts
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Condylomata Acuminata | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Intervention Model Description: Healthy women ages 20-45 eligible for the trial will be stratified at a 1: 1 ratio into 2 age subgroups (20-30 years of age and 31-45 years of age), and each subgroup will be randomized at a 1: 1: 1 ratio to receive the mid-dosage investigational vaccine, high-dosage investigational vaccine or the positive control, respectively.
Who Masked: Participant, Investigator
Masking Description: The Sponsor, investigators and biostatisticians will remain blinded to subject allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Group of Investigational Vaccine (Experimental): For Mid-dosage group, 0.5-mL suspension for injection, each 0.5-mL prefilled syringe dose contains L1 proteins of HPV types 6/11/16/18/31/33/45/52/58 in the amounts of 30μg#40μg#60μg#40μg#20μg#20μg#20μg#20μg and 20μg respectively, totaling 270μg of antigens.
  For High-dosage group, 0.5-mL suspension for injection, each 0.5-mL prefilled syringe dose contains L1 proteins of HPV types 6/11/16/18/31/33/45/52/58 in the amounts of 30μg#40μg#80μg#60μg#30μg#30μg#30μg#30μg and 30μg respectively, totaling 360μg of antigens.
  Interventions: Biological: Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli)
- The Group of Active Control Vaccine (Active Comparator): 0.5-mL suspension for injection, each 0.5-mL single-dose syringe contains approximately 20 mcg of HPV Type 6 L1 protein, 40 mcg of HPV Type 11 L1 protein, 40 mcg of HPV Type 16 L1 protein, 20 mcg of HPV Type 18 L1 protein, totaling 120 mcg of antigens.
  Interventions: Biological: Recombinant Quadrivalent Human Papillomavirus (Types 6,11,16,18) Vaccine (Saccharomyces cerevisiae)

INTERVENTIONS:
Biological: Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli) — For Mid-dosage group, a 3-dose regimen administered at months 0, 2 and 6.
  For High-dosage group, a 3-dose regimen administered at months 0, 2 and 6.
  Arms: The Group of Investigational Vaccine
Biological: Recombinant Quadrivalent Human Papillomavirus (Types 6,11,16,18) Vaccine (Saccharomyces cerevisiae) — A 3-dose regimen administered at months 0, 2 and 6.
  Arms: The Group of Active Control Vaccine

SUMMARY:
This trail is to evaluate the safety profile of Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli) in healthy Chinese women ages 20-45 and determine the optimal ratio of the antigens included in the investigational vaccine. Besides, the trail is also to demonstrate that the levels of neutralizing antibodies to vaccine HPV types 31, 33, 45, 52 and 58 elicited by the investigational vaccine with the chosen optimal antigen ratio are superior to those induced by Gardasil.

DETAILED DESCRIPTION:
This is a single-center, blinded, randomized and Gardasil-controlled (quadrivalent HPV vaccine GARDASIL®) Phase II clinical trial.

The trial will recruit a total of approximately 780 Chinese women 20-45 years of age with permanent residence. Healthy women ages 20-45 eligible for the trial will be stratified at a 1: 1 ratio into 2 age subgroups (20-30 years of age and 31-45 years of age), and each subgroup will be randomized at a 1: 1: 1 ratio to receive the mid-dosage investigational vaccine, high-dosage investigational vaccine or the positive control (quadrivalent HPV vaccine GARDASIL®), respectively.

Each subject will be administered 0.5 ml of the investigational vaccine or control in accordance with a 3-dose regimen at months 0, 2 and 6.

Peripheral blood samples of each subject will be collected at Day 0 (prior to dose 1), Month 7 (1 month post dose 3) to determine the levels of neutralizing antibodies and IgG antibodies to HPV types 6/11/16/18/31/33/45/52/58 in the sera. Optimal ratio of the antigens included in the investigational vaccine will be decided based on the immunogenicity and safety data from this trail.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects ages 20-45 (inclusive of 20 years of age and 45 years of age);
2. Subjects decided to be healthy by the principal investigator in accordance with such trial subjects' medical history and physical examination results;
3. Subjects who agree to participate in the trial after being fully informed of the study, and provide a written informed consent;
4. Trial subjects who are able to comply with protocol-specified requirements;
5. Trial subjects with negative urine pregnancy test at screening;
6. Trial subjects with no childbearing potential (e.g. females who have undergone bilateral tubal ligation, hysterectomy, bilateral oophorectomy, etc), or female subjects with childbearing potential who have agreed to abstain from any sexual activity that could result in pregnancy or practice adequate contraception for at least 28 days prior to the first dose of the interventions and throughout the study.
7. Subjects with axillary temperature≤37.0℃.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding, or planning for pregnancy in the following 7 months;
2. Women who have received other HPV vaccine(s) prior to dose 1 of the interventions;
3. Women who have received an investigational or unregistered drug or vaccine within 28 days prior to the first dose of the interventions, or plan to receive an investigational or unregistered drug or vaccine during the study;
4. Women who have known anaphylaxis history or are allergic to any component of the interventions, such as penicillin and amikacin;
5. Women with a history of severe adverse reactions to previous vaccinations, such as allergies, urticaria, dyspnea, angioneurotic edema, or abdominal pain;
6. Women who have an autoimmune disease or immunodeficiency, are HIV positive, or have primary diseases in vital organs;
7. Women who have asthma that is unstable and requires urgent care, hospitalization and the use of oral or intravenous corticosteroids during the past 2 years;
8. Women who have diabetes mellitus (type I or II), with the exception of gestational diabetes;
9. Women with a history of thyroidectomy or thyroid diseases that required medical care within the past 12 months;
10. Women with serious angioedema episodes within the past 3 years or requiring medical care over the past 2 years
11. Women who have hypertension over 145/95 at enrolment despite being treated by medication;
12. Women with coagulation disorders as diagnosed by a doctor (e.g. coagulation factor deficiency, coagulopathy, or platelet disorder) or coagulation difficulty
13. Women with active malignancy, or treated malignancy for which there is no reasonable assurance of sustained cure, or malignancy that is likely to recur during the study;
14. Women with epilepsy other than epilepsy with febrile seizures under the age of two, epilepsy secondary to alcohol use 3 years prior to alcohol withdrawal, or a singular epileptic seizure not requiring treatment within the past 3 years;
15. Women with the condition of asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen;
16. Women with a history of systematic chemotherapy in the past 5 years, a history of immunosuppressive therapy and cytotoxic therapy, and treatment with inhaled corticosteroids within the past 6 months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis);
17. Women who received blood products in the 3 months prior to vaccination with the interventions;
18. Women who received a live attenuated vaccine during the 28 days prior to vaccination with the interventions;
19. Women who received a subunit or inactivated vaccine, such as pneumococcal vaccine, or underwent antianaphylactic treatment during the 14 days prior to vaccination with the interventions;
20. Women who are currently on an anti-TB prophylaxis or therapy;
21. Women who had fever (with axillary temperature≥38.0℃) during the 3 days prior to vaccination with the interventions, or onset of any acute illness that required the use of antibiotics and antiviral treatment within the past 5 days;
22. Women with psychiatric conditions that preclude compliance with the protocol, or women with past or present psychoses, past or present bipolar disorder that has not been well controlled over the past 2 years, or women who are on medication for psychoses, or women who had suicidal thoughts/tendency in the past 5 years prior to enrolment;
23. Women with any medical, psychological or social conditions, or for occupational reasons or otherwise as judged by the principal investigator, that preclude participation in the study, or compromise such subject's ability to give informed consent.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 780 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Percentage of adverse reactions up to Day 7 after each dose of the interventions | 0-7 days after each immunization
  Percentage of subjects with 1 or more injection-site or non-injection-site (systemic) adverse reactions up to Day 7 after each dose of the interventions
To determine the optimal ratio of antigens included in the investigational vaccine | The 1st month after full immunization
  To determine the optimal ratio of antigens included in the investigational vaccine through non-inferiority analysis of the GMTs of neutralizing antibodies specific to vaccine HPV types 6, 11, 16 and 18 elicited by the investigational vaccine versus those induced by the positive control, in subjects negative for antibodies to such vaccine HPV types prior to dose 1.

SECONDARY OUTCOMES:
Percentage of adverse events up to Day 30 after each dose of the interventions | 0-30 days after each immunization
  Percentage of subjects with 1 or more injection-site or non-injection-site (systemic) adverse events up to Day 30 after each dose of the interventions
Percentage of erious adverse events for the duration of the study | Through study completion, an average of 7 months
  Percentage of subjects with serious adverse events for the duration of the study (from Day 1 till Month 7)
To demonstrate that the levels of neutralizing antibodies | The 1st month after full immunization
  To demonstrate that the levels of neutralizing antibodies specific to vaccine HPV types 31, 33, 45, 52 and 58 elicited by the investigational vaccine with the chosen optimal antigen ratio are superior to those induced by Gardasil through assessing the GMTs of neutralizing antibodies to HPV types 31, 33, 45, 52 and 58 in the sera of the subjects who are negative for antibodies to such HPV types prior to dose 1 of the investigational vaccine in comparison with those administered Gardasil.
To evaluate the levels of neutralizing antibodies | The 7th month after first immunization
  Subgroup Analysis: To evaluate the levels of neutralizing antibodies to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1.
To evaluate the levels of IgG antibodies | The 7th month after first immunization
  Subgroup Analysis: To evaluate the levels of IgG antibodies to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1.
To evaluate the rates of seropositivity | The 7th month after first immunization
  Subgroup Analysis: To evaluate the rates of seropositivity to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1.
To evaluate the rates of seroconversion | The 7th month after first immunization
  Subgroup Analysis: To evaluate the rates of seroconversion to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1.
To evaluate the levels of neutralizing antibodies among all subjects | The 7th month after first immunization
  To evaluate the levels of neutralizing antibodies to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among all subjects.
To evaluate the levels of IgG antibodies among all subjects | The 7th month after first immunization
  To evaluate the levels of IgG antibodies to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among all subjects.
To evaluate the rates of seropositivity among all subjects | The 7th month after first immunization
  To evaluate the rates of seropositivity to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among all subjects.
To evaluate the rates of seroconversion among all subjects | The 7th month after first immunization
  To evaluate the rates of seroconversion to each HPV type (HPV 6/11/16/18/31/33/45/52/58) at Month 7 post dose 1 among all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjiang Liu, Bachelor, Study Chair — Beijing Health Guard Biotechnology, Inc
Locations (1):
- CDC, Jiangsu Province, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
No informed consent was obtained to disclose the subject's data and sample test results

REFERENCES:
- [Derived] Wei M, Liu H, Yu H, Pan H, Tao H, Zhang J, Han W, Wu D, Wang W, Li J. Immunogenicity and safety of an Escherichia coli-produced 9-valent human papillomavirus vaccine (types 6/11/16/18/31/33/45/52/58) in healthy Chinese women aged 20-45 years: a single-center, randomized, observer-blinded, positive controlled phase 2 clinical trial. Front Immunol. 2025 Nov 14;16:1706662. doi: 10.3389/fimmu.2025.1706662. eCollection 2025. PMID 41322412